CLINICAL TRIAL: NCT04522128
Title: Does Quality of Life Decline During the COVID-19 Pandemic and Can we Change Behaviour to Improve Poor Quality of Life?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Tracy Epton, Lecturer, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2020-9463-15184
Record Dates: First submitted 2020-05-12; First posted 2020-08-21 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: COVID; Quality of Life; Behavior; Social Isolation
Keywords: COVID; Behaviour Change; Prevention; Quality of Life; Social Isolation
MeSH Terms: conditions — Behavior; Social Isolation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Feedback Intervention (Active Comparator): All participants will complete an online questionnaire. This will include demographic information, social distancing/isolation history, The Lubben Social Network Scale, The 6-item Loneliness Scale, Ten-Item Personality Scale, Spontaneous Self-affirmation Scale, Brief Illness Perception Questionnaire and the WHOQoL COMBI plus importance of QOL facet questions.
  Participants randomly allocated to the feedback intervention will then be provided with graphs showing WHOQOL COMBI facet scores and their perceived importance ratings. The graphs will highlight where quality of life might be poor but important to the participant. Participants will be asked three questions (i.e. how could your QoL in this domain be improved, what resources would you need to make this change, what practical actions are needed to address the discrepancies in your QoL?) to help them plan how they might be able to improve quality of life currently rated as poor but important.
  Interventions: Behavioral: Behaviour Change Technique Intervention to Improve Quality of Life
- Extended Intervention (Experimental): All participants will complete an online questionnaire (as described above).
  Participants randomly allocated to the extended intervention will then be provided with graphs to highlight differences between their actual WHOQoL COMBI scores and their perceived importance ratings. The graphs will highlight where quality of life might be poor but important to the participant. Participants will be asked three questions (i.e. how could your QoL in this domain be improved, what resources would you need to make this change, what practical actions are needed to address the discrepancies in your QoL?) to help them plan how they might be able to improve quality of life currently rated as poor but important.
  Participants will then receive an online intervention that will provide them with behaviour change techniques to help them address the discrepancies in the relevant quality of life domains.
  Interventions: Behavioral: Behaviour Change Technique Intervention to Improve Quality of Life
- Waitlist Control (Other): All participants will complete an online questionnaire. This will include demographic information, social distancing/isolation history, The Lubben Social Network Scale, The 6-item Loneliness Scale, Ten-Item Personality Scale, Spontaneous Self-affirmation Scale, Brief Illness Perception Questionnaire and the WHOQoL COMBI plus importance of QOL facet questions.
  Participants randomly allocated to the waitlist control group will then receive their WHOQoL COMBI scores only, with no information about differences between quality of life and importance or intervention materials.
  Interventions: Behavioral: Behaviour Change Technique Intervention to Improve Quality of Life

INTERVENTIONS:
Behavioral: Behaviour Change Technique Intervention to Improve Quality of Life — The intervention targets each facet of the five domains of WHOQOL COMBI. The intervention is based on the COM-B Framework (Michie et al., 2012) and utilises behaviour change techniques to help participants change their behaviour to improve their quality of life.
  The intervention will be compared to an active comparator 'feedback intervention' and a waitlist control group.

SUMMARY:
The response to COVID-19 means social isolation/distancing for the majority of the UK. This has the potential to negatively affect all domains of quality of life (QoL). QoL can be improved by giving feedback on gaps between someone's perceived QoL in a domain and how important it is to them (plus prompting reflective questions). However, interventions that are designed to improve QoL may increase the effectiveness of this as optimised behaviour change techniques can be used. This study aims to develop and test a quality of life intervention during social isolation/distancing.

DETAILED DESCRIPTION:
The response to COVID-19 means social isolation/distancing for the majority of the UK. This has the potential to negatively affect all domains of quality of life (QoL). QoL can be improved by giving feedback on gaps between someone's perceived QoL in a domain and how important it is to them (plus prompting reflective questions). However, interventions that are designed to improve QoL may increase the effectiveness of this as optimised behaviour change techniques can be used. This study aims to develop and test a quality of life intervention during social isolation/distancing.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18+ years
* Living in United Kingdom during COVID-19 pandemic.

Exclusion Criteria:

* English language - all participants are required to be able to read and understand English to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Change in World Health Organisation Quality of Life Combination | Change from baseline quality of life to 2 weeks post intervention
  Measure of quality of life, score ranges from 0-100 per domain, with a higher score indicating greater quality of life
Change in World Health Organisation Quality of Life Combination | Change from baseline quality of life to 3 months post intervention
  Measure of quality of life, score ranges from 0-100 per domain, with a higher score
Change in World Health Organisation Quality of Life Combination | Change from baseline quality of life to 6 months post intervention
  Measure of quality of life, score ranges from 0-100 per domain, with a higher score

SECONDARY OUTCOMES:
Change in The Lubben Social Network Scale | Change from baseline social isolation to 2 weeks post intervention
  Measure of social isolation, score ranges between 0 and 30, with a higher score indicating more social engagement.
Change in The Lubben Social Network Scale | Change from baseline social isolation to 3 months post intervention
  Measure of social isolation, score ranges between 0 and 30, with a higher score indicating more social engagement.
Change in The Lubben Social Network Scale | Change from baseline social isolation to 6 months post intervention
  Measure of social isolation, score ranges between 0 and 30, with a higher score indicating more social engagement.
Change in 6-Item Loneliness Scale | Change from baseline loneliness to 2 weeks post intervention
  Measure of loneliness, score ranges between 0 and 50, with a higher score indicating less loneliness.
Change in 6-Item Loneliness Scale | Change from baseline loneliness to 3 months post intervention
  Measure of loneliness, score ranges between 0 and 50, with a higher score indicating less loneliness.
Change in 6-Item Loneliness Scale | Change from baseline loneliness to 6 months post intervention
  Measure of loneliness, score ranges between 0 and 50, with a higher score indicating less loneliness.
Quality of Life Importance Ratings | Change from baseline importance to 2 weeks post intervention
  Measure of importance of different facets of quality of life, score ranges 0-200, with a higher score indicating greater importance of quality of life.
Quality of Life Importance Ratings | Change from baseline importance to 3 months post intervention
  Measure of importance of different facets of quality of life, score ranges 0-200, with a higher score indicating greater importance of quality of life.
Quality of Life Importance Ratings | Change from baseline importance to 6 months post intervention
  Measure of importance of different facets of quality of life, score ranges 0-200, with a higher score indicating greater importance of quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Epton, Principal Investigator — University of Manchester
Locations (1):
- University of Manchester - online, Manchester, Cheshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
WHOQOL COMBI data cannot be shared with researchers outside of the research team.